CLINICAL TRIAL: NCT07340944
Title: Comparison of the Effects of N-acetylcysteine, Calcium Hydroxide, and Double Antibiotic Paste on Postoperative Pain Level, Periapical RANKL/OPG Ratio, and Antibacterial Activity
Brief Title: Comparison of the Effects of N-acetylcysteine, Calcium Hydroxide, and Double Antibiotic Paste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ceren Yeniay, PhD, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU-DF-CY-01
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Apical Periodontitis
Keywords: N-acetylcysteine; calcium hydroxide; double antibiotic paste; intracanal medicament; RANKL; osteoprotegerin; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetylcysteine; Calcium Hydroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- N-acetylcysteine group (Experimental): NAC was placed into the root canal as an intracanal medication.
  Interventions: Drug: N Acetyl Cysteine
- Calcium Hydroxide Group (Active Comparator): Ca(OH)2 was placed into the root canal as an intracanal medication.
  Interventions: Drug: Calcium Hydroxide (Ca(OH)2)
- Double Antibiotic Paste Group (Active Comparator): DAP was placed into the root canal as an intracanal medication.
  Interventions: Drug: Double Antibiotic Paste

INTERVENTIONS:
Drug: N Acetyl Cysteine — NAC was placed into the root canal as an intracanal medication. The medication was removed after one week. Root canal treatment was completed. Treatment was completed for 15 patients in the group within one month.
  Arms: N-acetylcysteine group
Drug: Calcium Hydroxide (Ca(OH)2) — Ca(OH)2 was placed into the root canal as an intracanal medication. The medication was removed after one week. Root canal treatment was completed. Treatment was completed for 15 patients in the group within one month.
  Arms: Calcium Hydroxide Group
Drug: Double Antibiotic Paste — DAP was placed into the root canal as an intracanal medication. The medication was removed after one week. Root canal treatment was completed. Treatment was completed for 15 patients in the group within one month.
  Arms: Double Antibiotic Paste Group

SUMMARY:
This study aimed to evaluate the efficacy of N-acetylcysteine (NAC) used as an intracanal medicament on antibacterial activity, periapical RANKL/OPG ratio, and postoperative pain levels.

DETAILED DESCRIPTION:
Apical periodontitis (AP) is a condition characterized by a dominant inflammatory response in the root canal system of the affected tooth and irreversible inflammation of the periradicular tissues caused by a microbial infection . Endodontic treatment is considered the gold standard treatment for apical periodontitis because it completely removes the pulp tissue and biofilm. During this process, lesions that may occur in the periradicular tissues due to endodontic origin can be minimized, reduced, or completely eliminated .

Numerous irrigation protocols and intracanal medications, including various mechanical instrumentation techniques, have been developed to reduce microorganisms and inflammation in the root canal system and to control pain . Intracanal medications are antibacterial agents placed within the root canal between sessions to eliminate residual microorganisms . These medications exhibit anti-inflammatory effects, thereby reducing pain, eliminating apical exudate, controlling inflammatory root resorption, and preventing contamination between sessions . However, numerous published articles on endodontic infection control debate the effectiveness of existing intracanal drugs These conflicting findings complicate the determination of an ideal intracanal drug for endodontic treatments and have led researchers to search for more effective and reliable alternatives.

N-acetylcysteine (NAC), a sulfhydryl group-containing compound with mucolytic properties, was first patented in 1960 and began to be used in medicine in 1967 . In recent years, it has been evaluated as a potential agent as an irrigating solution and intracanal medicament in endodontics. Numerous in vitro studies on the antimicrobial activity of NAC have demonstrated its high antimicrobial activity against planktonic microorganisms and multispecies biofilms responsible for endodontic infections, including Enterococcus faecalis . In addition to inhibiting the production and release of proinflammatory cytokines , it is a potent thiol-containing antioxidant with high antimicrobial activity. Furthermore, one of the limited clinical studies on the use of NAC as an intracanal medication reported significantly increased levels of the pro-resolving lipid mediators RvE1 and RvD2 in the periapical tissues of teeth treated with NAC as an intracanal medication, whereas a similar increase was not observed in the calcium hydroxide (Ca(OH)₂)-treated group . These findings demonstrate that NAC is not only noteworthy for its antimicrobial activity but also for its biological properties that may contribute to the resolution of the inflammatory response.Antimicrobial activity alone is not sufficient to assess the clinical efficacy of intracanal medicaments; the biological effects of these agents on periapical tissues should also be considered. In this context, the Nuclear factor kappa-B receptor activator ligand (RANKL)/Osteoprotegerin (OPG) ratio, a key indicator of osteoclastic activity, is a valuable biomarker for biochemically assessing treatment response in endodontic treatments because it reflects the effect of inflammation on bone destruction. Increasing RANKL levels and decreasing OPG levels have been associated with root-end resorption and periapical lesion progression. Furthermore, postoperative pain, which directly impacts patients' quality of life, is one of the key criteria for evaluating the clinical success of intracanal medications. Therefore, this study aimed to conduct a holistic analysis of intracanal medicaments from both biological and clinical perspectives by evaluating not only antimicrobial activity but also the RANKL/OPG ratio and postoperative pain levels.

To date, there are no randomized controlled trials using NAC as an intracanal medication, where each of its antibacterial activity, RANKL/OPG ratio, and effect on postoperative pain levels has been clinically evaluated. This study, which is the first to examine these three parameters separately at the clinical level, aims to evaluate the effects of NAC on postoperative pain, antibacterial activity, and the RANKL/OPG ratio by comparing it with Ca(OH)₂ and double antibiotic paste (DAP). For this purpose, our study aims to test the null hypothesis that NAC, Ca(OH)₂, and DAP used as intracanal medications have no effect on antibacterial activity, RANKL/OPG ratio, or postoperative pain levels.

ELIGIBILITY:
Inclusion Criteria:

* Non-vital teeth confirmed by clinical and pulp sensitivity tests
* Teeth with a single canal and diagnosed with asymptomatic apical periodontitis
* Periapical assessment (PAI) of 2 or greater
* Teeth with a pocket depth not exceeding 3 mm
* Teeth without excessive root curvature (Schneider class 1) and with visible root canals on radiographs
* Permanent teeth with complete root development
* Patients between the ages of 18 and 65
* Teeth without previous endodontic treatment

Exclusion Criteria:

* Patients who refused to participate in the study
* Patients with any systemic disease
* Patients who received antibiotic treatment within the last 3 months
* Patients who were pregnant or suspected of being pregnant
* Teeth with excessive crown damage that would not allow for the placement of a rubber dam
* Teeth with root fractures, pathological findings or mobility,
* Presence of any resorption in the involved tooth,
* Patients with active swelling and tenderness to palpation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Antibacterial efficacy of intracanal medicaments, RANKL/OPG ratio and effect on postoperative pain | The medication will remain in the canal for one week. Patients will receive treatment within one month.
  The antibacterial activity of intracanal medicaments will be measured by PCR analysis, Rankl/opg ratio will be measured by ELISA analysis and postoperative level will be measured by VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Yeniay, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No